CLINICAL TRIAL: NCT02918188
Title: Therapeutic Effects of Hydrogen on Steroid-refractory/or Steroid-dependent Chronic Graft-versus-host-disease
Brief Title: Therapeutic Effects of Hydrogen on Steroid-refractory/or Steroid-dependent cGVHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Doctor, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NavyGHB-004
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Chronic Graft-versus-host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Hydrogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrogen (Experimental): Patients will receive hydrogen-rich water (4mL/kg three times one day, 0.8 ppm)
  Interventions: Drug: Hydrogen

INTERVENTIONS:
Drug: Hydrogen — Patients will receive hydrogen-rich water orally (500mL three times one day, 0.6mM)
  Other Names: Hydrogen-rich water

SUMMARY:
This study suggested that hydrogen has a potential as an effective and safe therapeutic agent on cGVHD.

DETAILED DESCRIPTION:
The investigators will evaluate clinical response rate, time to treatment Failure (TTF), overall survival (OS), and toxicity in cGVHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male
* not pregnant female
* patients <65 years old
* Diagnosis of cGVHD steroid refractory (no response after Prednisone ≥1mg/kg ) or steroid-dependent cGVHD (had an initial response followed by a cGVHD flare upon steroid taper)
* Patient intolerant to steroid therapy

Exclusion Criteria:

* Patients with stable disease, not well controlled by the current treatment
* Pregnancy
* HIV positive
* Severe liver or renal impairment: serum creatinine >2.5 mg/dl; serum bilirubin>2.5 mg/dl (without evidence of hepatic cGVHD)
* Uncontrolled malignancies including the persistence of the underlying malignancy before the Allogeneic Transplantation and the relapse of hematopoietic malignancy
* Any other investigational agents administered within last four weeks
* Cardiac insufficiency (>grade II, New York Heart Association classification)
* Inability to comply with medical therapy or follow-up

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 12 months after date of start of Hydrogen
  Overall Response Rate (ORR) is defined as an Objective improvement at sixth month, and includes at least 1 of the following criteria:
  At least 50% reduction of body surface area involved; Reduction (at least 20%) of skin sclerosis, measured by Rodnan score Improvement>1 point in functional pulmonary tests, evaluated by LFS score; >50% steroid reduction (for at least 4 weeks)

SECONDARY OUTCOMES:
Response Rate in each domain (RRD) | 12 months after date of start of Hydrogen
  Response rate in each domain was measured in subjects that had had initial involvement in that domain

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, M.D., Study Chair — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian L, Liu M, Shen J, Cen J, Zhao D. Hydrogen in Patients With Corticosteroid-Refractory/Dependent Chronic Graft-Versus-Host-Disease: A Single-Arm, Multicenter, Open-Label, Phase 2 Trial. Front Immunol. 2020 Nov 25;11:598359. doi: 10.3389/fimmu.2020.598359. eCollection 2020. PMID 33324415